CLINICAL TRIAL: NCT06394622
Title: A Clinical Research About CD70-targeted CAR-NKT Cells Therapy Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Head of Phase I Clinical Trial Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGC729-IIT-02
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cyclophosphamide + Fludarabine + Infusion of CAR-NKT Cells (Experimental): Lymphodepleting regimen, Cyclophosphamide 250mg/m2 IV on day -5 to -3 and Fludarabine 25mg/m2 IV on days -5 to -3. Followed by infusion of CAR-NKT on day 0.
  Potential CGC729 doses:
  Dose level 1: 5.0×106 CAR- NKT cells/m2; Dose level 2: 1.5×107 CAR- NKT cells/m2;
  Interventions: Combination Product: Cyclophosphamide + Fludarabine + Infusion of CAR-NKT Cells

INTERVENTIONS:
Combination Product: Cyclophosphamide + Fludarabine + Infusion of CAR-NKT Cells — Biological: CD70 CAR-NKT cells. Drug: Cyclophosphamide. Drug: Fludarabine.

SUMMARY:
This is a phase I, open-label, single-arm study conducted to evaluate the efficacy, safety and PK of CGC729 in the treatment of advanced malignant solid tumors.

Condition or disease:advanced malignant solid tumors. Intervention/treatment:Biological: CD70 CAR-NKT cells. Phase:I

DETAILED DESCRIPTION:
This was a dose-expansion study, we plan to enroll 6 to 12 patients with CD70-positive advanced malignant solid tumors to CGC729 treatment. The intended enrollment for the evaluation of treatment efficacy and safety was planned to be 3 to 6 patients per tumor type.

We used leukapheresis for cell collection. The lymphodepletion procedure was conducted using a combination of fludarabine and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years.
* ECOG 0-1 points.
* The expected survival time is more than 3 months.
* Patients with advanced advanced malignant solid tumor confirmed by histology or cytology to be recurrent or metastatic after at least second-line treatment.
* IHC: CD70 positive.
* At least one measurable lesion at baseline per RECIST version 1.1.
* The functions of important organs are basically normal:Hematopoietic function:

neutrophils 1.5×109/L, platelets 75×109/L, hemoglobin 80g/L;Renal function: creatinine clearance of ≥60 mL/min.;Liver function: ALT and AST ≤2.5×ULN (≤5 × ULN for patients with liver metastases);Total bilirubin ≤1.5×ULN.Prothrombin time (PT) : INR < 1.7.

* Pregnancy tests for women of childbearing age shall be negative, Both men and women agreed to use effective contraception.
* Subjects or their guardians agree to participate in this clinical trial and sign the ICF, indicating that they understand the purpose and procedures of this clinical trial and are willing to participate in the research.

Exclusion Criteria:

* Use of cell therapy within the previous one month.
* Risk of severe bleeding in esophageal cancer
* Subjects with other malignant tumors within the past 2 years, except basal or squamous skin cancer, superficial bladder cancer, and breast cancer in situ, have been completely cured and do not need follow-up treatment.
* Patients with leptomeningeal metastasis or central nervous system metastasis, and definite central nervous system underlying diseases with significant symptoms in the past 6 months.
* Immunotherapy, targeted drug therapy or chemotherapy within 5 drug half-lives within 2 weeks before cell infusion.
* Active hepatitis B, HIV positive and HCV positive
* Active infection or uncontrollable infection.
* Subjects with NYHA heart failure class ≥2 or hypertension uncontrolled by standard therapy requiring special treatment, previous history of myocarditis, or myocardial infarction within 6 months.
* Unstable respiratory diseases, including interstitial pneumonia.
* Uncontrolled ascites and pleural effusion
* Known to have active or uncontrolled autoimmune diseases, such as Crohns disease, rheumatoid arthritis, systemic lupus erythematosus, etc. .
* Subjects who are using systemic steroids or steroid inhalers for treatment.
* Pregnant or lactating female subjects.
* Other investigators deem it unsuitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
ORR of CD70 CAR-NKT cell dynamics | Day 1 through week 56
  Assess Objective response rate

SECONDARY OUTCOMES:
DCR of CD70 CAR-NKT cell dynamics | Day 1 through week 56
  Disease control rate
DOR of CD70 CAR-NKT cell dynamics | Day 1 through week 56
  Duration of Response
PFS of CD70 CAR-NKT cell dynamics | Day 1 through week 56
  Progress Free Survival
OS of CD70 CAR-NKT cell dynamics | Day 1 through week 56
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Principal Investigator — Fudan University
Locations (1):
- Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No